CLINICAL TRIAL: NCT05526950
Title: Cytokine Filtration in Lung Transplantation - a Randomised, Controlled, Multicentre Clinical Trial (GLUSorb)
Brief Title: Cytokine Filtration in Lung Transplantation: A Swedish National Study (GLUSorb)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Principal Investigator, Sandra Lindstedt, Professor, Lund University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLUSorb
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Lung Transplant Failure; Lung Transplant; Complications

STUDY DESIGN:
Intervention Model Description: The model consists of a randomized controlled in human patients using a "cytokine adsorption" device.
  Lung transplant recipients are randomized to either the treatment group which undergoes cytokine adsorption using the medical device compared to the control group which has not received the cytokine adsorber.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated (Active Comparator): Treatment using the medical "cytokine adsorption" device in conjunction with lung transplantation
  Interventions: Device: Device: CytoSorb
- Non-treated (No Intervention): No additional treatment in conjunction with lung transplantation

INTERVENTIONS:
Device: Device: CytoSorb — Medical device used hemoperfusion and cytokine adsorption in conjunction with lung transplantation.
  Arms: Treated

SUMMARY:
Lung transplantation (LTx) remains the gold standard for treating patients with irreversible end-stage pulmonary disease. Of the major organs transplanted, survival in LTx recipients remains the lowest (mean 5 years). Despite improvements, primary graft dysfunction (PGD), as defined by respiratory insufficiency and edema up to 72 hours post LTx, remains the leading cause of early mortality and contributes to the development of chronic lung allograft dysfunction (CLAD) which is the leading cause of late mortality. PGD develops within the first 72 hours after LTx. The development of CLAD increases quickly with cumulative incidence of 40-80 % within the first 3-5 years. There is a general lack of efficient treatments for PGD and CLAD. Prevention of PGD is therefore of crucial importance and has a direct impact on survival.

The present study is a randomized controlled study which aims to compare patients undergoing LTx with and without the utilization of cytokine adsorption.

DETAILED DESCRIPTION:
Early intolerance to the newly transplanted lung starts at the time of transplantation and results in PGD driven by an intense inflammatory response. Cytokines play a critical role as signaling molecules that initiate, amplify, and maintain inflammatory responses both locally and systemically. The use of cytokine filtration devices to target middle- and low-molecular weight molecules has been shown to reduce levels of a diverse number of cytokines. These results have been demonstrated in the in vitro reduction of pathogen-associated molecular pattern molecules (PAMPS) and damage associated molecular patterns (DAMPS) as well as in in vivo studies involving orthotopic heart transplantation and kidney transplantation. Cytokine adsorption has been used successfully in clinical applications to both heart and kidney transplantation.

The present study is a randomized controlled study which aims to collect preliminary data on the efficacy of a medical device through the comparison of patients undergoing LTx with and without cytokine adsorption.

ELIGIBILITY:
Inclusion Criteria:

• Eligibility to undergo double lung transplantation at either trial site

Exclusion Criteria:

1. Age <18 years
2. Previous organ transplantation
3. Presence of any conditions at the time of surgery that require immunosuppressive therapy. Immunosuppressive therapy is defined as:

   1. Cyclosporine, Tacrolimus, Everolimus, or Sirolimus, minimum 1 month of treatment prior to transplantation and active treatment at the time of transplantation.
   2. Any form of antibody-based treatment that is known for having an immunomodulatory effect taken up to 1 week before transplantation.
4. Non-consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine whether cytokine reduction by cytokine filtration leads to improved oxygenation in patients undergoing lung transplantation. | First 72 hours after lung transplantation
  Higest value of oxygenation expressed as the PaO2/FiO2 ratio.
To determine whether cytokine reduction by cytokine filtration leads to improved oxygenation in patients undergoing lung transplantation. Oxygenation at 24 hours | 24 hours after lung transplantation
  Oxygenation expressed as the PaO2/FiO2 ratio at 24 hours
To determine whether cytokine reduction by cytokine filtration leads to improved oxygenation in patients undergoing lung transplantation. Oxygenation at 48 hours | 48 hours after lung transplantation
  Oxygenation expressed as the PaO2/FiO2 ratio at 48 hours
To determine whether cytokine reduction by cytokine filtration leads to improved oxygenation in patients undergoing lung transplantation. Oxygenation at 72 hours | 72 hours after lung transplantation
  Oxygenation expressed as the PaO2/FiO2 ratio at 72 hours

SECONDARY OUTCOMES:
To determine whether cytokine reduction by cytokine filtration improves levels of plasma inflammatory markers (including cytokines) in patients undergoing lung transplantation. | 0-72 hours (0-3 days) after lung transplantation
  Plasma levels of inflammatory markers: interleukin (IL)-10, IL-1β, soluble IL-2 receptor, IL-6, IL-8, and tumour necrosis factor (TNF)α before and immediately after transplantation and at 6, 12, 24, 48, and 72 hours after transplantation, and C-reactive protein (CRP) and white blood cells before and immediately after transplantation and at day 1, 2, and 3 after transplantation
To determine whether cytokine reduction by cytokine filtration decreases lung infiltrates and oedema in patients undergoing lung transplantation | 0-72 hours (0-3 days) after lung transplantation
  Infiltrates and oedema measured by chest x-ray and/or CT scan of the thorax at day 1, 2, and 3 after transplantation
To determine whether cytokine reduction by cytokine filtration improves arterial blood gas measures in patients undergoing lung transplantation | 0-72 hours (0-3 days) after lung transplantation
  Highest daily arterial blood gas measurements recorded on day 1, 2, and 3 after transplantation, as a measure of lung function
To determine whether cytokine reduction by cytokine filtration decreases severity of primary graft dysfunction (PGD) in patients undergoing lung transplantation | 0-72 hours (0-3 days) after lung transplantation
  PGD severity as evaluated per standard clinical procedures using a rating scale from 0-3 on day 1, 2, and 3 after transplantation, as a measure of lung function
To determine whether cytokine reduction by cytokine filtration decreases incidence of primary graft dysfunction (PGD) in patients undergoing lung transplantation | 0-72 hours (0-3 days) after lung transplantation
  Presence of any grade of PGD on day 1, 2, and 3 after transplantation, as a measure of lung function
To determine whether cytokine reduction by cytokine filtration decreases need for norepinephrine in patients undergoing lung transplantation | 0-72 hours (0-3 days) after lung transplantation
  Total dose of norepinephrine administered in the first 72 h
To determine whether cytokine reduction by cytokine filtration decreases mortality in patients undergoing lung transplantation | First 4 years
  Mortality up to 48 months after transplantation
To determine whether cytokine reduction by cytokine filtration improves diffusion capacity of the lungs (DLCO) in patients undergoing lung transplantation | First 4 years
  Lung diffusion capacity, measured by carbon monoxide (CO) diffusion, at 6, 12, 24, and 48 months after transplantation, as a measure of lung function
To determine whether cytokine reduction by cytokine filtration improves forced expiratory volume (FEV1), forced vital capacity (FVC), and total lung capacity in patients undergoing lung transplantation | First 4 years
  Forced expiratory volume (FEV1), forced vital capacity (FVC), and total lung capacity (TLC) measured by spirometry at 1, 3, 6, 12, 24 and 48 months after transplantation, as a measure of lung function
To determine whether cytokine reduction by cytokine filtration improves occurrence of any acute rejection episodes in patients undergoing lung transplantation | First 4 years
  Occurrence of any acute rejection episodes (clinically treated and/or biopsy verified) up to 48 months after transplantation, as a measure of lung function
To determine whether cytokine reduction by cytokine filtration improves Chest CT in patients undergoing lung transplantation | First 4 years
  Chest CT findings at 1, 3, 6, 12, 24, 36 and 48 months after transplantation
To determine whether cytokine reduction by cytokine filtration improves presence of any CLAD in patients undergoing lung transplantation | First 4 years
  Presence of any CLAD and CLAD subtypes up to 48 months after transplantation, as a measure of lung function
To determine whether cytokine reduction by cytokine filtration improves kidney function in patients undergoing lung transplantation | First 4 years
  Kidney function evaluated by measurement of serum creatinine levels; calculated glomerular filtration rate (GFR); and need for renal replacement therapy on day 1, 2, and 3 and at 1, 3, 6, 9, 12, 24, and 48 months after transplantation; urea levels on day 1, 2, and 3 after transplantation; and iohexol clearance at 3, 6, 9, 12, 24, 36, and 48 months after transplantation
To determine whether cytokine reduction by cytokine filtration improves quality of life (QOL) in patients undergoing lung transplantation | First 4 years
  QOL evaluated by the 36-Item Short Form Health Survey (SF-36) at 24 and 48 months after transplantation

OTHER OUTCOMES:
Safety endpoints | First 72 hours after transplantation
  Adverse events in the first 72 hours after transplantation. Thus, the aim of this clinical trial is to determine the efficacy of cytokine filtration in improving successful LTx rates, based on its effects on oxygenation ratio, pulmonary function, PGD, kidney function, CLAD, and survival. These outcomes will also be analysed on the molecular, and tissue levels to identify the mechanisms by which cytokine filtration promotes the acceptance of lung transplants. The primary outcome will be oxygenation ratio, defined as the highest PaO2/FiO2 (P/F) within 72 h after LTx.
Exploratory endpoints | First 4 years
  Collection of a portion of routinely collected transplanted lung tissue by transbronchial biopsy and bronchoalveolar lavage fluid (at least at 1, 3 and 12 months, with additional timepoints if clinically indicated), collection of explanted recipient lung tissue, and collection of blood samples (at least before transplantation; immediately after transplantation; 6, 12, 24, 48, and 72 hours; 1 and 2 weeks; and 1, 3, 6, 9, 12, 24, 36, and 48 months after transplantation, with additional timepoints if clinically indicated) in a biobank for future exploratory analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Lindstedt, MD, PhD, Principal Investigator — Skånes universitetssjukhus Lund
Locations (1):
- Sandra Lindstedt, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No
All results will be presented at group level. No individual data.

REFERENCES:
- [Background] Ghaidan H, Stenlo M, Niroomand A, Mittendorfer M, Hirdman G, Gvazava N, Edstrom D, Silva IAN, Broberg E, Hallgren O, Olm F, Wagner DE, Pierre L, Hyllen S, Lindstedt S. Reduction of primary graft dysfunction using cytokine adsorption during organ preservation and after lung transplantation. Nat Commun. 2022 Jul 26;13(1):4173. doi: 10.1038/s41467-022-31811-5. PMID 35882835
- [Background] Niroomand A, Qvarnstrom S, Stenlo M, Malmsjo M, Ingemansson R, Hyllen S, Lindstedt S. The role of mechanical ventilation in primary graft dysfunction in the postoperative lung transplant recipient: A single center study and literature review. Acta Anaesthesiol Scand. 2022 Apr;66(4):483-496. doi: 10.1111/aas.14025. Epub 2022 Jan 27. PMID 35014027
- [Background] Niroomand A, Hirdman G, Olm F, Lindstedt S. Current Status and Future Perspectives on Machine Perfusion: A Treatment Platform to Restore and Regenerate Injured Lungs Using Cell and Cytokine Adsorption Therapy. Cells. 2021 Dec 29;11(1):91. doi: 10.3390/cells11010091. PMID 35011653
- [Background] Lindstedt S, Niroomand A, Mittendorfer M, Hirdman G, Hyllen S, Pierre L, Olm F. Nothing but NETs: Cytokine adsorption correlates with lower circulating nucleosomes and is associated with decreased primary graft dysfunction. J Heart Lung Transplant. 2023 Oct;42(10):1358-1362. doi: 10.1016/j.healun.2023.06.011. Epub 2023 Jun 20. PMID 37348689
- [Derived] Lindstedt S, Silverborn M, Lannemyr L, Pierre L, Larsson H, Grins E, Hyllen S, Dellgren G, Magnusson J. Design and Rationale of Cytokine Filtration in Lung Transplantation (GLUSorb): Protocol for a Multicenter Clinical Randomized Controlled Trial. JMIR Res Protoc. 2023 Dec 13;12:e52553. doi: 10.2196/52553. PMID 37855706